CLINICAL TRIAL: NCT03420092
Title: A Randomized, 6-period, 6-treatment, Single-dose, Open-label, Single-center, Crossover Study to Assess the Relative Bioavailability of Different Formulations of AZD5718 and the Food Effect on the Selected Formulation of AZD5718 in Healthy Volunteers
Brief Title: A Study to Assess the Bioavailability of Different Formulations of AZD5718 and the Food Effect on the Selected Formulation of AZD5718 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D7550C00005
Record Dates: First submitted 2018-01-18; First posted 2018-02-05 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Coronary Artery Disease
Keywords: vasoactive leukotrienes by leukocytes; bioavailability
MeSH Terms: conditions — Coronary Artery Disease | interventions — AZD5718

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Treatment A (Experimental): The participant will be administered with Form 1 of AZD5718 tablets with an overnight fast of at least 10 hours.
  Interventions: Drug: Form 1 of AZD5718 tablets
- Treatment B (Experimental): The participant will be administered with Form 2 of AZD5718 tablets with an overnight fast of at least 10 hours.
  Interventions: Drug: Form 2 of AZD5718 tablets
- Treatment C (Experimental): The participant will be administered with Form 3 of AZD5718 tablets with an overnight fast of at least 10 hours.
  Interventions: Drug: Form 3 of AZD5718 tablets
- Treatment D (Experimental): The participant will be administered with Form 4 of AZD5718 tablets with an overnight fast of at least 10 hours.
  Interventions: Drug: Form 4 of AZD5718 tablets
- Treatment E (Experimental): The participant will be administered with Form 5 of AZD5718 tablets with an overnight fast of at least 10 hours.
  Interventions: Drug: Form 5 of AZD5718 tablets
- Treatment F (Experimental): The participant will be administered with selected form (one of Form 2-5) of AZD5718 tablets 30 minutes after start of the meal.
  Interventions: Drug: Selected form (Form 2 - 5) of AZD5718 tablets

INTERVENTIONS:
Drug: Form 1 of AZD5718 tablets — The participants will be dosed with Form 1 of AZD5718 following an overnight fast of at least 10 hours.
  Arms: Treatment A
Drug: Form 2 of AZD5718 tablets — The participants will be dosed with Form 2 of AZD5718 following an overnight fast of at least 10 hours.
  Arms: Treatment B
Drug: Form 3 of AZD5718 tablets — The participants will be dosed with Form 3 of AZD5718 following an overnight fast of at least 10 hours.
  Arms: Treatment C
Drug: Form 4 of AZD5718 tablets — The participants will be dosed with Form 4 of AZD5718 following an overnight fast of at least 10 hours.
  Arms: Treatment D
Drug: Form 5 of AZD5718 tablets — The participants will be dosed with Form 5 of AZD5718 following an overnight fast of at least 10 hours.
  Arms: Treatment E
Drug: Selected form (Form 2 - 5) of AZD5718 tablets — The participant will be administered with selected form (one of Form 2-5) of AZD5718 tablets 30 minutes after start of the meal.
  Arms: Treatment F

SUMMARY:
In this study, the relative bioavailability of different formulations of AZD5718 will be determined in order to compare it with the formulation used in a previous Phase 2a study and confirm appropriate drug exposure. This study consist of 2 parts. In Part 1, 5 different formulations of AZD5718 would be provided to the participant in fasting condition in a randomized order. After evaluation of Part 1 a single formulation would be selected for dosing in fed condition in Part 2. Each participant will be involved in the study for approximately 5 to 6 weeks. Fourteen participants will be randomized to ensure at least 10 evaluable participants at the end of the last treatment period.

DETAILED DESCRIPTION:
This is a Randomized, 6-period, 6-treatment, Single-dose, Open-label, Single-center, Crossover, phase I Study to Assess the Relative Bioavailability of Different Formulations of AZD5718 and the Food Effect on the Selected Formulation of AZD5718 in Healthy Volunteers. In this study, the relative bioavailability of different formulations of AZD5718 will be determined in order to compare it with the formulation used in a previous Phase 2a study and confirm appropriate drug exposure. The optimal pharmacokinetic (PK) profile of AZD5718 is currently not known but working hypothesis is that a flatter PK profile will deliver the same efficacy at a lower dose/exposure compared to a fluctuating AZD5718 profile. Thus, formulations with different release rates will be evaluated. Potential food effect of a selected formulation would be determined in order to provide appropriate dose and dosing instructions for further development of AZD5718. This study would consist of 2 parts. In Part 1, 5 different formulations of AZD5718 would be provided to the participants in fasting condition in a randomized order. After evaluation of Part 1 a single formulation would be selected for dosing in fed condition in Part 2. Part 1 of the study will be an open-label, randomized, 5-period, 5-treatment, single dose crossover study in 14 healthy participants (males and females of non-childbearing potential), performed at a single study center to ensure that at least 10 participants are evaluable. Each participant would be randomized to 1 of 10 treatment sequence according to a Williams design to receive the 5 treatments as following: Form 1 of AZD5718 tablets, Treatment B: Form 2 of AZD5718 tablets, Treatment C: Form 3 of AZD5718 tablets, Treatment D: Form 4 of AZD5718 tablets, and Treatment E: Form 5 of AZD5718 tablets. Participants will receive 1 treatment per treatment period. During each treatment period, participants would be dosed following an overnight fast of at least 10 hours. No fluids will be allowed apart from water which can be given until 2 hours before administration of the investigational medicinal product (IMP) and then from 1 hours after administration of the IMP. The dose would be administered with 240 mL of water. A standard meal would be given 4 hours after administration of the IMP. Participants should not lie fully supine (unless specified for certain assessments) for 4 hours after dosing. After completion the PK evaluation in Part 1, the formulation for Part 2 would be selected. At least 10 participants from Part 1 will be included in Part 2, to ensure that at least 8 participants are evaluable. For each participant included in Part 2, there would be minimum period of at least 2 weeks between the last dose of IMP in Part 1 and the dose of IMP in Part 2. During the treatment period in Part 2, participants would be dosed with the selected formulation of IMP with food. Participants would fast at least 10 hours prior to receiving the test meal. Participants should start the recommended meal 30 minutes prior to administration of the IMP. Participants would be required to consume the meal in 25 minutes; however, the IMP should be administered 30 minutes after start of the meal with 240 mL of water. No fluids would be allowed apart from water which can be given until 1 hour before administration of the IMP and then from 2 hours after administration of the IMP. Each participant will be involved in the study for approximately 5 to 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent before any study specific procedures.
2. Healthy male and/or female subjects aged 18 to 55 years (inclusive) with suitable veins for cannulation or repeated venipuncture.
3. Females must have a negative pregnancy test at screening and on admission to the unit, must not be lactating and must be of non childbearing potential, confirmed at screening by fulfilling one of the following criteria 3.1. Postmenopausal defined as amenorrhoea for at least 12 months or more following cessation of all exogenous hormonal treatments and follicle stimulating hormone (FSH) levels in the postmenopausal range.

   3.2. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
4. Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
5. Provision of signed, written and dated informed consent for optional genetic/biomarker research. If a subject declines to participate in the genetic component of the study, there will be no penalty or loss of benefit to the subject. The subject will not be excluded from other aspects of the study described in this protocol.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the PI, may either put the volunteer at-risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
2. History or presence of gastrointestinal (GI), hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
3. Participants with any special dietary restrictions such as subjects that are lactose intolerant or are vegetarians/vegans.
4. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
5. Any clinically significant abnormalities in clinical chemistry, hematology or urinalysis results, at screening and/or admission to the study unit as judged by the PI.
6. Any clinically significant abnormal findings in vital signs at screening, as judged by the PI.
7. Any clinically significant abnormalities on 12-lead ECG at screening and/or admission to the study unit, as judged by the PI.
8. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.
9. Known of suspected Gilbert's syndrome and known or suspected history of drug abuse, as judged by the PI.
10. Has received another new chemical or biological entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study. The period of exclusion begins 3 months after the final dose or one month after the last visit whichever is the longest.

    Note: Participants consented and screened, but not randomized in this study or a previous phase I study, are not excluded.
11. Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months before screening.
12. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the PI or history of hypersensitivity to drugs with a similar chemical structure or class to AZD5718.
13. Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the 3 months before screening.
14. Positive screen for drugs of abuse or cotinine (screening only) at screening or on each admission to the study center or positive screen for alcohol on each admission to the study center.
15. Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks before the first administration of IMP.
16. Use of any prescribed or non prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks before the first administration of IMP or longer if the medication has a long half life.
17. Known or suspected history of alcohol or drug abuse or excessive intake of alcohol as judged by the PI.
18. Involvement of any AstraZeneca, PAREXEL or study site employee or their close relatives.
19. Subjects who have previously received AZD5718.
20. Judgment by the PI that the subject should not participate in the study if they have any ongoing or recent minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements.
21. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship.
22. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection or previous bone marrow transplant.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve (AUC) of AZD5718 | At pre dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36 and 48 hours post dose.
  To assess the pharmacokinetics (PK) parameter AUC to evaluate the relative bioavailability of different formulations of AZD5718 and compare with the formulation (Form 1 of AZD5718 tablets) used in the Phase 2a clinical study.
AUC from time zero to time of last quantifiable concentration (AUC[0-t]) of AZD5718 | At pre dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36 and 48 hours post dose.
  To assess the PK parameter AUC(0-t)to evaluate the relative bioavailability of different formulations of AZD5718 and compare with the formulation (Form 1 of AZD5718 tablets) used in the Phase 2a clinical study.
Observed maximum plasma concentration (Cmax) of AZD5718 | At pre dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36 and 48 hours post dose.
  To assess the PK parameter Cmax to evaluate the relative bioavailability of different formulations of AZD5718 and compare with the formulation (Form 1 of AZD5718 tablets) used in the Phase 2a clinical study.
Observed plasma concentration at 24 hours post dose (C24) of AZD5718 | 24 hour post dose
  To assess the PK parameter C24 to evaluate the relative bioavailability of different formulations of AZD5718 and compare with the formulation (Form 1 of AZD5718 tablets) used in the Phase 2a clinical study.

SECONDARY OUTCOMES:
Cmax of AZD5718 in fed and fasted conditions | At pre dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36 and 48 hours post dose.
  To assess the ratio of Cmax of a selected AZD5718 formulation when administered in fed and fasted conditions and relative bioavailability of the tested formulations.
C24 of AZD5718 in fed and fasted conditions | At pre dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36 and 48 hours post dose.
  To assess the ratio of C24 of a selected AZD5718 formulation when administered in fed and fasted conditions and relative bioavailability of the tested formulations.
AUC(0-t) of AZD5718 in fed and fasted conditions | At pre dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36 and 48 hours post dose.
  To assess the ratio of AUC(0-t) of a selected AZD5718 formulation when administered in fed and fasted conditions and relative bioavailability of the tested formulations.
AUC of AZD5718 in fed and fasted conditions | At pre dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36 and 48 hours post dose.
  To assess the ratio of AUC of a selected AZD5718 formulation when administered in fed and fasted conditions and relative bioavailability of the tested formulations.
Number of participants with adverse events | From randomization throughout the treatment period (Day 1 to 3) and follow-up Visit (Day 5 to 7) assessed maximum upto 6 weeks.
  All adverse events will be coded using MedDRA vocabulary, and will be listed for each subject.
Assessment of systolic blood pressure | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose].
  To assess the systolic blood pressure as a criteria of safety and tolerability.
Assessment of diastolic blood pressure | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose].
  To assess the Diastolic blood pressure as a criteria of safety and tolerability.
Assessment of pulse rate | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose].
  To assess Pulse rate as a criteria of safety and tolerability.
Assessment of 12-lead electrocardiogram (ECG) | At screening (From Day -28 to Day -2 - Part 1); 5 to 7 days post final dose (Part 2).
  To assess the ECG as a criteria of safety and tolerability. A 10 second 12 lead ECG will be obtained after 10 minutes supine rest.
Assessment of physical examination | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose].
  Assessment of physical examinations will include an assessment of the general appearance, respiratory, cardiovascular, abdomen, skin, head, and neck (including ears, eyes, nose, and throat), lymph nodes, thyroid, musculoskeletal and neurological systems.
Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve (t½λz) of AZD5718 | At pre dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36 and 48 hours post dose.
  To assess PK parameter t½λz to evaluate the relative bioavailability of different formulations of AZD5718 and compare with the formulation (Form 1 of AZD5718 tablets) used in the Phase 2a clinical study.
Time to reach maximum observed plasma concentration (Tmax) of AZD5718 | At pre dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36 and 48 hours post dose.
  To assess the PK parameter Tmax to evaluate the relative bioavailability of different formulations of AZD5718 and compare with the formulation (Form 1 of AZD5718 tablets) used in the Phase 2a clinical study.
Apparent total body clearance of drug from plasma after extravascular administration (CL/F) of AZD5718 | At pre dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36 and 48 hours post dose.
  To assess the PK parameter CL/F to evaluate the relative bioavailability of different formulations of AZD5718 and compare with the formulation (Form 1 of AZD5718 tablets) used in the Phase 2a clinical study.
Safety and tolerability of AZD5718 by assessment of clinical Laboratory evaluations (Hematology)- white blood cell (WBC) count | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of WBC count.
Safety and tolerability of AZD5718 by assessment of clinical Laboratory evaluations (hematology)- red blood cell (RBC) count | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of RBC count.
Safety and tolerability of AZD5718 by assessment of clinical Laboratory evaluations (hematology)- haemoglobin (HB) | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of HB.
Safety and tolerability of AZD5718 by assessment of clinical Laboratory evaluations (hematology)- hematocrit (HCT) | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of HCT.
Safety and tolerability of AZD5718 by assessment of clinical Laboratory evaluations (hematology)- platelets | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of platelets.
Safety and tolerability of AZD5718 by assessment of clinical Laboratory evaluations (hematology)- reticulocytes absolute count | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of reticulocytes absolute count.
Safety and tolerability of AZD5718 by assessment of clinical Laboratory evaluations (hematology)- mean corpuscular hemoglobin (MCH) | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of MCH.
Safety and tolerability of AZD5718 by assessment of clinical Laboratory evaluations (hematology)- mean corpuscular hemoglobin concentration (MCHC) | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of MCHC.
Safety and tolerability of AZD5718 by assessment of clinical laboratory evaluations (clinical chemistry)- creatinine | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of creatinine.
Safety and tolerability of AZD5718 by assessment of clinical laboratory evaluations (clinical chemistry)- creatine kinase | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of creatine kinase.
Safety and tolerability of AZD5718 by assessment of clinical laboratory evaluations (clinical chemistry)- total bilirubin | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of total bilirubin.
Safety and tolerability of AZD5718 by assessment of clinical laboratory evaluations (clinical chemistry)- unconjugated bilirubin | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of unconjugated bilirubin.
Safety and tolerability of AZD5718 by assessment of clinical laboratory evaluations (clinical chemistry)- alkaline phosphatase | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of alkaline phosphatase.
Safety and tolerability of AZD5718 by assessment of clinical laboratory evaluations (clinical chemistry)- aspartate aminotransferase (AST) | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of AST.
Safety and tolerability of AZD5718 by assessment of clinical laboratory evaluations (clinical chemistry)- gamma glutamyl transpeptidase (GGT) | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of GGT.
Safety and tolerability of AZD5718 by assessment of clinical laboratory evaluations (clinical chemistry)- albumin | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of albumin.
Safety and tolerability of AZD5718 by assessment of clinical laboratory evaluations (clinical chemistry)- potassium | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of potassium.
Safety and tolerability of AZD5718 by assessment of clinical laboratory evaluations (clinical chemistry)- sodium | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of sodium.
Safety and tolerability of AZD5718 by assessment of clinical Laboratory evaluations (clinical chemistry)- calcium | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of calcium.
Safety and tolerability of AZD5718 by assessment of clinical laboratory evaluations (clinical chemistry)- C-reactive protein | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of C-reactive protein.
Safety and tolerability of AZD5718 by assessment of clinical Laboratory evaluations (clinical chemistry)- urea | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of urea.
Safety and tolerability of AZD5718 by assessment of clinical laboratory evaluations (clinical chemistry)- phosphate | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of phosphate.
Safety and tolerability of AZD5718 by assessment of clinical laboratory evaluations (clinical chemistry)- glucose (fasting) | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of glucose (fasting).
Safety and tolerability of AZD5718 by assessment of clinical laboratory evaluations- urinalysis (blood) | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of urinalysis (blood). If urinalysis is positive for blood, a microscopy test will be performed to assess RBC, white blood cell [WBC], casts [cellular, granular, hyaline]).
Safety and tolerability of AZD5718 by assessment of clinical laboratory evaluations- urinalysis (glucose) | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of urinalysis (glucose).
Safety and tolerability of AZD5718 by assessment of clinical laboratory evaluations (hematology)- Mean corpuscular volume (MCV) | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of MCV.
Safety and tolerability of AZD5718 by assessment of clinical laboratory evaluations (clinical chemistry)- Alanine aminotransferase (ALT) | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of ALT
Safety and tolerability of AZD5718 by assessment of clinical laboratory evaluations (clinical chemistry)- Thyroxine 4 (T4) | At screening (From Day -28 to Day-2)
  Safety and tolerability of AZD5718 by assessment of T4.
Safety and tolerability of AZD5718 by assessment of clinical laboratory evaluations(clinical chemistry)- Thyroid stimulating hormone (TSH) | At screening (From Day -28 to Day-2)
  Safety and tolerability of AZD5718 by assessment of TSH.
Safety and tolerability of AZD5718 by assessment of clinical laboratory evaluations(clinical chemistry)- Follicle stimulating hormone (FSH) | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of FSH in female participants.
Safety and tolerability of AZD5718 by assessment of clinical laboratory evaluations (hematology)- Neutrophils absolute count | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of neutrophils absolute count.
Safety and tolerability of AZD5718 by assessment of clinical laboratory evaluations (hematology)- Lymphocytes absolute count | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of lymphocytes absolute count.
Safety and tolerability of AZD5718 by assessment of clinical laboratory evaluations (hematology)- Monocytes absolute count | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of monocytes absolute count.
Safety and tolerability of AZD5718 by assessment of clinical laboratory evaluations (hematology)- Basophils absolute count | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of basophils absolute count.
Safety and tolerability of AZD5718 by assessment of clinical laboratory evaluations- urinalysis (protein) | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of urinalysis (protein). If urinalysis is positive for protein, a microscopy test will be performed to assess RBC, WBC, casts [cellular, granular, hyaline]).
Safety and tolerability of AZD5718 by assessment of clinical laboratory evaluations (hematology)- Eosinophils absolute count | [Part 1 - At screening (From Day -28 to Day-2); Treatment period 1 (Day-1), Treatment period 1 to 5 (Day 1 to 3)] and [Part 2- At Day-1, Day 1 to 3, 5 to 7 days post final dose]
  Safety and tolerability of AZD5718 by assessment of eosinophils absolute count.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Forte Soto, MD, Principal Investigator — PAREXEL Early Phase Clinical Unit London
Locations (1):
- Research Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided